CLINICAL TRIAL: NCT04519827
Title: A Prospective, Randomised, Double-blind Controlled Study, to Evaluate the Safety/Hypoallergenicity of a New Rice-based Hydrolysate Formula With New Ingredient for Infants and Children With Diagnosed Cow's Milk Allergy
Brief Title: A Hypoallergenicity Study on a New Rice-Based Hydrolysate Formula
Acronym: CHARM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Schär AG / SPA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CHARM-01-2020
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Allergy;Food
Keywords: Cow's Milk Protein Allergy (CMPA); Cow's Milk Allergy (CMA); CHILDREN
MeSH Terms: conditions — Food Hypersensitivity; Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New Rice-based hydrolysate (Experimental): The TEST formula is a new Rice-based hydrolysate with new ingredient.
  Interventions: Other: New Rice-based hydrolysate
- Amino-acid based formula (Placebo Comparator): The PLACEBO is an Amino-acid based formula.
  Interventions: Other: Amino Acid-based infant formula

INTERVENTIONS:
Other: New Rice-based hydrolysate — A rice-based hydrolysed infant formula with new ingredient
  Arms: New Rice-based hydrolysate
Other: Amino Acid-based infant formula — An amino acid-based infant formula
  Arms: Amino-acid based formula

SUMMARY:
Cow's Milk Allergy (CMA) affects between 2-3% of young children but its severity varies between regions/countries. While the long-term prognosis for CMA is good, with the majority (80-90%) of children outgrowing their allergy by around 3-5 years. Breast feeding is the most optimal form of feeding for all infants, regardless of their condition, and in those with CMA maternal dairy exclusion is recommended as first line treatment. In non-breast fed or mixed feeding, a hypoallergenic milk substitute is recommended for young infants. The AAP and other societies such as EAACI and ESPGHAN considers a formula to be 'hypoallergenic' if at least 90% of children with documented CMA tolerate it, with a 95% CI, under double-blind, placebo-controlled conditions.This equates to at least 29 children who should tolerate the product following blind and open challenge.

DETAILED DESCRIPTION:
A prospective, multi-centre double blind randomised placebo-controlled study to demonstrate the safety and tolerance of a new rice-based hydrolysate in children with diagnosed Cow's Milk Allergy (CMA). The test product being a new milk substitute hydrolysed rice-based formula with new ingredient. The results will satisfy the safety requirement when tolerated by 90% of children with proven CMA, with a confidence of 95%. New, and previously diagnosed children with confirmed CMA who meet the inclusion criteria will be eligible to participate in the study. Those included in the intervention phase will have IgE testing and an oral food challenge (OFC) to test and placebo products, in a randomised double-blind design. Children with a negative reaction to both test and placebo products will receive the test product for a period of 7 days (open challenge).

ELIGIBILITY:
Inclusion Criteria:

1. Children <10 yrs of age
2. Proven IgE-mediated CMA
3. >2500g at birth
4. > 37 weeks gestation
5. Written informed consent provided by parent(s)/guardian

Exclusion Criteria:

1. Infants/children with severe concurrent illness (other than food allergy/CMA)
2. Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements.
3. Participation in other studies involving use of milk replacement products designed to treat/manage CMA within two weeks prior to entry into this study
4. Current participation in OIT to Cow's Milk
5. Diagnosis of anaphylaxis to Cow's Milk
6. Diagnosis of rice allergy

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Hypoallergenicity | 7 days open challenge
  90% of children tolerate the TEST formula with a 95% CI - using the double blind placebo controlled food challenge and open challenge (Test vs. placebo).

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (3):
  - Meyer Children's Hospital, Florence
  - Spett.le Universita degli Studi di Napoli ''Federico II'', Napoli
  - Hospital Infantile Regina Margherita., Turin
- Hospital Sant Joan de Déu Barcelona 2020,, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No